CLINICAL TRIAL: NCT05896696
Title: Prospective Clinical Study for the Evaluation of the Efficacy and Safety of the BeShape One Device for Non-invasive Waist Circumference Reduction
Brief Title: Efficacy and Safety of the BeShape One Device for Non-invasive Waist Circumference Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BeShape Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-BSO-001
Record Dates: First submitted 2023-05-17; First posted 2023-06-09 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Dermatological Non-Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BeShape One Device Treatment (Experimental)
  Interventions: Device: BeShape One

INTERVENTIONS:
Device: BeShape One — Single treatment with the BeShape One device. Participants will receive treatment on at least 4 abdomen/flanks treatment areas and up to 6 treatment areas, at the discretion of the investigator. The subject will receive one treatment on each treatment area.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of the BeShape One device for non-invasive waist circumference reduction in adults between the ages of 18 and 65. The main question[s] it aims to answer are:

* reduction in waist circumference following treatment with the BeShape One device at the final 6 and 12-week follow-up visits compared to baseline
* Subject improvement and satisfaction
* Investigator satisfaction
* Subject comfort/pain level

Participants will undergo a single treatment with the BeShape One device at the Baseline visit and will return for two follow up visits at 6 and 12 weeks post treatment.

Researchers will compare the results at the follow up visits to Baseline.

DETAILED DESCRIPTION:
This study is a prospective, baseline controlled, multi-center, one arm clinical study aimed to assess the efficacy and safety of the BeShape OneTM device for waist circumference reduction.

Seventy (70) subjects in two investigational sites will be enrolled in this study. All subjects will undergo an assessment of their general health. A single treatment utilizing the BeShape OneTM device will be administered.

During the follow-up period, visits will be conducted as follows: 6 weeks (6wk FU), and 12 weeks (12wk FU) post treatment. Subject's waist circumference will be measured at baseline (before treatment) and at each of the follow up visits. Circumference reduction will be assessed at each post baseline visit, using a standardized and validated measuring technique. Additionally, investigator and subject assessments will be completed at each follow up visit. Photography of the treatment areas will be performed under visible light conditions of the front, right, left and back view of the subjects at the baseline visit (before first treatment) and at the last follow-up visit (12wk FU).

ELIGIBILITY:
Inclusion Criteria:

1. Female and male subjects ≥18 and ≤65 years of age.
2. Abdominal fat thickness of at least 1.5 cm (measured by calibrated caliper).
3. 18.5 ≤ BMI ≤ 33
4. Women of childbearing potential (i.e., not post-menopausal or surgically sterilize) must have a negative urine pregnancy test. Participating women of childbearing potential must be using a medically acceptable form of birth control for at least 3 months prior to enrollment.
5. Understand the study and volunteer to sign the informed consent.
6. Willing to follow the treatment and follow up schedule and post-treatment care instructions.
7. Willing to refrain from a change in diet, exercise or medication regimen for the duration of the study.
8. Willing to have de-identified images of the treated areas taken for possible use in publications and presentations.

Exclusion Criteria:

1. Pregnant women, intending to become pregnant during the study, less than 12 months after delivery, breastfeeding, or less than 6 weeks after completing breastfeeding;
2. Participation in another clinical study of another investigational device or drug involving the same anatomical site within the last 3 months, or, if it does not involve the same anatomical site, at the discretion of the researcher.
3. Subjects with significant systemic disease, such as ongoing hyperlipidemia, diabetes mellitus, hepatitis or other liver disease, HIV-positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease, and malignant neoplasms; undergoing chronic steroid or immunosuppressive therapy.
4. Subject having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
5. An implanted pacemaker or any other implantable active device anywhere in the body.
6. Subjects with thyroid disease and / or metabolic syndrome.
7. Unstable weight within the last 6 months (i.e. + 3% weight change in the past six months).
8. Local skin pathologies or natural structure loss in the treated area (hernia) and / or loss of sensation or dysesthesia in the treated area.
9. Previous body contouring procedures in the treatment area within the past 12 months.
10. History of abdominal surgery, including laparoscopic procedures.
11. Caesarean section within 12 months.
12. Any permanent or temporary implant in the treatment area such as metal plates or an injected chemical substance such as silicone.
13. Actively expressed psychiatric or psychological state.
14. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months.
15. Any condition that, at the researcher's discretion, renders the subject unsuitable for participation in a clinical research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahava Stein, Study Director — A. Stein Regulatory Affairs Consulting Ltd.
Locations (2):
- Chicago Cosmetic Surgery and Dermatology, Chicago, Illinois, United States
- Centro Poliklinika, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BeShape One Device Treatment
Started | 81
Completed | 72
Not Completed | 9
Not completed — Screening Failure | 7
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | BeShape One Device Treatment
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.29 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 67
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42
  Lithuania | 30
Height [Mean (Standard Deviation); unit: cm] | 169.4 (10.12)
Weight [Mean (Standard Deviation); unit: kg] | 74.6 (12.71)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (2.88)
Waist circumference [Mean (Standard Deviation); unit: cm] | 90.3 (9.44)

OUTCOME MEASURES:

1. Primary Outcome: Change in Waist Circumference
Description: Waist circumference change (in cm) following BeShape treatment at the final 12 week follow-up visit compared to baseline.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | BeShape One Device Treatment
Number analyzed (Participants) | 72
cm | -1.87 (2.62)
Statistical Analysis 1: Comparison: BeShape One Device Treatment; Test type: Other; p < 0.0001, Paired sample t-test; Mean Difference (Final Values) = -1.87, 95% CI 2-sided [-2.49 to -1.26]

2. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference change (in cm) following BeShape treatment at the 6 week follow up visits compared to baseline.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | BeShape One Device Treatment
Number analyzed (Participants) | 72
cm | -1.22 (2.06)
Statistical Analysis 1: Comparison: BeShape One Device Treatment; Test type: Other; p < 0.0001, paired sample t-test; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-1.70 to -0.73]

3. Secondary Outcome: Subject Improvement
Description: Subject improvement is measured using the Global Aesthetic Improvement (GAI) scale at each follow up visit. The GAI scale is a 7 point scale ranging from significantly worse (-3) to significant improvement (+3). A higher GAI score indicates a greater improvement.
Time Frame: 6 and 12 weeks
Population: Five (5) participants did not complete the 6 weeks follow-up (FU) visit and seven (7) participants did not complete their 12 weeks FU visit. Reasons for not completing the follow up visits: 4 participants were lost to follow up (2 did not return for the 6 and 12 week FU visit and 2 did not return only for the 12 week FU visit), 1 participant became pregnant after the treatment and was dropped from the study and 2 participants did not complete the treatment and therefore did not return for FU
Measure: Count of Participants; unit: Participants
Arm/Group | BeShape One Device Treatment
Number analyzed (Participants) | 67
Participants
  6 weeks: (3) Very much improved (significant improvement) | 3
  6 weeks: (2) Much improved (moderate improvement) | 8
  6 weeks: (1) Improved (slight improvement) | 27
  6 weeks: (0) No change | 27
  6 weeks: (-1) Worse (slightly worse) | 2
  6 weeks: (-2) Moderately Worse | 0
  6 weeks: (-3) Significantly Worse | 0
  12 weeks: number analyzed (Participants) | 65
  12 weeks: (3) Very much improved (significant improvement) | 2
  12 weeks: (2) Much improved (moderate improvement) | 5
  12 weeks: (1) Improved (slight improvement) | 29
  12 weeks: (0) No change | 28
  12 weeks: (-1) Worse (slightly worse) | 1
  12 weeks: (-2) Moderately Worse | 0
  12 weeks: (-3) Significantly Worse | 0

4. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction is measured using a 5 point Likert scale at each follow up visit. The 5 point Likert scale ranges from very dissatisfied (-2) to very satisfied (+2). A higher score indicates greater subject satisfaction.
Time Frame: 6 and 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BeShape One Device Treatment
Number analyzed (Participants) | 67
Participants
  6 weeks: (2) Very satisfied | 9
  6 weeks: 1) Satisfied | 27
  6 weeks: (0) No opinion | 25
  6 weeks: (-1) Dissatisfied | 6
  6 weeks: (-2) Very dissatisfied | 0
  12 weeks: number analyzed (Participants) | 65
  12 weeks: (2) Very satisfied | 2
  12 weeks: 1) Satisfied | 27
  12 weeks: (0) No opinion | 30
  12 weeks: (-1) Dissatisfied | 6
  12 weeks: (-2) Very dissatisfied | 0

5. Secondary Outcome: Investigator Satisfaction
Description: Investigator satisfaction is measuring using the Clinical Global Aesthetic Improvement (CGAI) scale at each follow up visit. The CGAI scale is a 7 point scale ranging from significantly worse (-3) to significant improvement (+3). A higher CGAI score indicates a greater improvement.
Time Frame: 6 and 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | BeShape One Device Treatment
Number analyzed (Participants) | 67
Participants
  6 weeks: (3) Very much improved (significant improvement) | 2
  6 weeks: (2) Much improved (moderate improvement) | 17
  6 weeks: (1) Improved (slight improvement) | 29
  6 weeks: (0) No change | 16
  6 weeks: (-1) Worse (slightly worse) | 3
  6 weeks: (-2) Moderately Worse | 0
  6 weeks: (-3) Significantly Worse | 0
  12 weeks: number analyzed (Participants) | 65
  12 weeks: (3) Very much improved (significant improvement) | 2
  12 weeks: (2) Much improved (moderate improvement) | 12
  12 weeks: (1) Improved (slight improvement) | 33
  12 weeks: (0) No change | 17
  12 weeks: (-1) Worse (slightly worse) | 1
  12 weeks: (-2) Moderately Worse | 0
  12 weeks: (-3) Significantly Worse | 0

6. Secondary Outcome: Subject Comfort/Pain
Description: Subject comfort/pain level will be assessed immediately after treatment using the Numeric Pain Rating Scale (NPRS). The NPRS scale is a 10 point scale ranging from 0 (no pain) to 10 (worst possible pain). A higher NPRS score indicates a greater pain level.
Time Frame: Immediately after the treatment procedure at Baseline, up to 5 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BeShape One Device Treatment
Number analyzed (Participants) | 72
score on a scale | 5.14 (1.73)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | BeShape One Device Treatment
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 1/72
Other Adverse Events (participants affected / at risk) | 47/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BeShape One Device Treatment (N=72)
Laparoscopically assisted hysterectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BeShape One Device Treatment (N=72)
Nasopharyngitis (Infections and infestations) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Uterine leiomyoma (Reproductive system and breast disorders) | 1 (1)
Application site bruise / Purpura (Skin and subcutaneous tissue disorders) | 11 (11)
Erythema (Skin and subcutaneous tissue disorders) | 34 (36)
Hyperaesthesia (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Edema (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may not publish the results of the Study, based on information collected or generated by Institution and Principal Investigator without the Sponsor's prior written consent. No publication, presentation in any forum or any other form of disclosure with respect to the Study or the results thereof will be made without Sponsor's prior written consent. The provisions shall apply during the term of the Agreement and for an additional period of 15 years following Study Completion.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT05896696/Prot_SAP_001.pdf